CLINICAL TRIAL: NCT04333927
Title: Adjuvant Immunotherapy Combined With Chemoradiation for Patients With High-risk reseCtable Extrahepatic chOlangiocaRcinoma and gallblaDder Cancer: a Phase II, Multicenter, Randomized Controlled Trial
Brief Title: Adjuvant Immunotherapy Combined With Chemoradiation for Patients With High-risk reseCtable Extrahepatic chOlangiocaRcinoma and gallblaDder Cancer
Acronym: ACCORD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTC001
Record Dates: First submitted 2020-04-02; First posted 2020-04-03 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Biliary Tract Cancer; Extrahepatic Cholangiocarcinoma; Gallbladder Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Drug Therapy; Observation; Immunotherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patients in treatment group will receive camrelizumab 200mg intravenously every 3 weeks until clinical or radiographic disease progression, unacceptable toxicity, death, termination of the study or withdrawal. After 1 or 2 courses of camrelizumab, patients went on to receive capecitabine (1,330 mg/m2 per day, in divided doses twice daily, 7 days per week) concurrent with radiotherapy (45 Gy to regional lymph nodes and 54 to 59.4 Gy to preoperative tumor bed).
  Interventions: Drug: Chemotherapy; Procedure: Immunotherapy; Radiation: Radiotherapy
- Observation (Placebo Comparator): Patients in observation group will not receive any anti-cancer therapy.
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Chemotherapy — Capecitabine (1,330 mg/m2 per day, in divided doses twice daily, 7 days per week).
  Arms: Treatment
Other: Observation — Patients in observation group will not receive any anti-cancer therapy.
  Arms: Observation
Procedure: Immunotherapy — Camrelizumab 200mg intravenously every 3 weeks until clinical or radiographic disease progression, unacceptable toxicity, death, termination of the study or withdrawal.
  Arms: Treatment
Radiation: Radiotherapy — 45 Gy to regional lymph nodes and 54 to 59.4 Gy to preoperative tumor bed.
  Arms: Treatment

SUMMARY:
The study is a multicenter phase II randomized controlled trial. The purpose is to investigate the efficacy and safety of adjuvant immunotherapy combined with chemoradiation for patients with high-risk resectable extrahepatic cholangiocarcinoma and gallbladder cancer.

DETAILED DESCRIPTION:
The trial will recruit 92 patients, and they will be randomized (1:1) into two groups (chemoradiation+immunotherapy group, observation group) after operation. Patients in chemoradiation+immunotherapy group will receive camrelizumab 200mg intravenously every 3 weeks until clinical or radiographic disease progression, unacceptable toxicity, death, termination of the study or withdrawal. After 1 or 2 courses of camrelizumab, patients went on to receive capecitabine (1,330 mg/m2 per day, in divided doses twice daily, 7 days per week) concurrent with radiotherapy (45 Gy to regional lymph nodes and 54 to 59.4 Gy to preoperative tumor bed). Patients in observation group will not receive any anti-cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years;
2. Primary resectable extrahepatic cholangiocarcinoma and gallbladder cancer proved by pathology which underwent radical surgery;
3. Pathology indicates R0 with T2-4 or N1; or R1;
4. ECOG PS 0-1;
5. Adequate hematologic, hepatic and renal function: ANC ≥ 1.5x10^9/L, Hb ≥ 80g/L, PLT ≥ 100 x10^9/L, albumin ≥ 28g/L, total bilirubin < 1.5×ULN, ALT and AST < 2.5×ULN, CREA<1.5×ULN;
6. At least 6 months of life expectancy.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or expecting to conceive or father children within the projected duration of the trial;
2. Received previous anti-cancer therapies;
3. With purulent, infected or delayed healed wounds;
4. Have risky bleeding events requiring transfusion, operation or local therapies, continuous medication in the past 3 months;
5. Have thromboembolism in the past 6 months, including myocardial infarction, unstable angina, stroke or transient ischemic attack, pulmonary embolism, deep vein thrombosis;
6. Have taken aspirin (>325mg/day) or other antiplatelet drugs continuously for 10 days or more within 2 weeks before enrolment;
7. Uncontrollable hypertension, systolic pressure>140mmHg or diastolic pressure>90mmHg after best medical care, or history of hypertensive crisis or hypertensive encephalopathy;
8. Symptomatic congestive heart failure (NYHA class II-IV). Symptomatic or badly-controlled arrhythmia. Congenital long QT syndrome or modified QTc>500ms upon screening;
9. Have active autoimmune diseases that require systemic treatment within 2 years before enrolment;
10. Active tuberculosis, having antituberculosis therapy at present or within 1 year;
11. Have a known history of prior invasive malignancies within 5 years before enrolment;
12. Have other uncontrollable comorbidities;
13. Infection of HIV, known syphilis requiring treatment;
14. Allergic to chemotherapeutics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | two years
  defined as the time from randomization until death from any cause. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive. Patients remaining alive throughout the duration of the study will have their survival time censored on the date last seen alive.

SECONDARY OUTCOMES:
Recurrence-free Survival | two years
  defined as the time from randomization until disease recurrence or death from any cause, whichever happens first. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive and recurrence-free. Patients not having an event will be censored at the date last seen alive.
Adverse Events | two years
  adverse events during the treatment period using Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, PhD, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xiao H, Ji J, Li S, Lai J, Wei G, Wu J, Chen W, Xie W, Wang S, Qiao L, Tu J, Shen S, Peng Z. Adjuvant Chemoradiation and Immunotherapy for Extrahepatic Cholangiocarcinoma and Gallbladder Cancer: A Randomized Clinical Trial. JAMA Oncol. 2025 Sep 1;11(9):1021-1029. doi: 10.1001/jamaoncol.2025.1926. PMID 40638104